CLINICAL TRIAL: NCT06718387
Title: Evaluation of the Impact of Participation in a Psycho-education Program for Victims of Sexual Violence
Acronym: PE-VVS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR-BDX-AP 2023-08
Record Dates: First submitted 2024-11-29; First posted 2024-12-05 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Ptsd; Sexual Violence; Therapeutic Alliance
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without group intervention (No Intervention): Patient refusing group care and/or assessment ended after the inclusion end dates
- With group intervention (Experimental): Patient in agreement with group management and available for participation
  Interventions: Other: PsychoEducation Program

INTERVENTIONS:
Other: PsychoEducation Program — 6 sessions of PsychoEducational Program
  Arms: With group intervention

SUMMARY:
Evaluation of the impact of a psycho-education program for victims of sexual violence, to determine the most efficient model to patients.

DETAILED DESCRIPTION:
In 2022, CRP Sud NA set up a psycho-education group for victims of sexual violence (PE-VVS). Two groups were held, involving 10 patients:

* Average age = 35 (29-50)
* Average PCL5 before PE-VSS = 53 (31 - 63)
* Type of SV experienced

  * In childhood or adolescence outside family environment
  * Incest
  * Rape in adulthood outside intimate relationship
  * Rape by intimate partner A special feature of this therapeutic group is the involvment of the CRP's patient-partner. He took part in both design and facilitation of the sessions, along with the two CRP co-therapists (IDE / psychologist).

ELIGIBILITY:
Inclusion Criteria:

* At the suggestion of CRP therapists,
* Patient treated at the CRP having been exposed to sexual violence

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of impact on quality of life (QoL) concerning participation in this psychoeducation program | 6 months after the end of program
  QoL measurement by Stages of Recovery Instrument "STORI"
Evaluation of impact on self-esteem of participation in this psychoeducation program | 6 months after the end of program
  Self-esteem measurement by Rosenberg self-esteem scale
Evaluation of Impact on mental well-being of participation in this psychoeducation program | 6 months after the end of program
  Well-being evalutation by Warwick-Edinburgh scale (WEMWBS)

CONTACTS AND LOCATIONS:
Overall Officials: Chantal BERGEY, Principal Investigator — Charles Perrens
Locations (1):
- Centre Hospitalier Charles PERRENS, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Millon EM, Shors TJ. Taking neurogenesis out of the lab and into the world with MAP Train My Brain. Behav Brain Res. 2019 Dec 30;376:112154. doi: 10.1016/j.bbr.2019.112154. Epub 2019 Aug 14. PMID 31421141
- [Background] Shors TJ, Millon EM. Sexual trauma and the female brain. Front Neuroendocrinol. 2016 Apr;41:87-98. doi: 10.1016/j.yfrne.2016.04.001. Epub 2016 Apr 13. PMID 27085856
- [Background] Shors TJ, Olson RL, Bates ME, Selby EA, Alderman BL. Mental and Physical (MAP) Training: a neurogenesis-inspired intervention that enhances health in humans. Neurobiol Learn Mem. 2014 Nov;115:3-9. doi: 10.1016/j.nlm.2014.08.012. Epub 2014 Sep 9. PMID 25219804